CLINICAL TRIAL: NCT02011984
Title: Multicentric Non-randomized Investigation of RESISTANT Camouflage Stent-system in Peripheral Superficial Femoral Arteries
Brief Title: Multicentric Non-randomized Investigation of RESISTANT Camouflage Stent-system
Acronym: RECAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eucatech AG (Industry)
Responsible Party: Sponsor
Other Study IDs: recam2013_eucatech; ECT024ResiCSfaRegV10 (Other: CERES)
Record Dates: First submitted 2013-11-15; First posted 2013-12-16 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- peripheral artery disease: de novo stenotic lesions in superficial femoral artery

SUMMARY:
Non-randomized multicenter post-market study to confirm the long-term safety and effectiveness of the CE-approved Camouflage-coated self-expandable RESISTANT Camouflage stent system for revascularization of de novo stenotic lesions in the superficial femoral artery in 100 compliant patients suitable for stent angioplasty.

The CE-approved device will be used according to its intended use. Beyond the standard of care no further interventions are scheduled. Therefore, this trial is subject to the exception to the rule §23b of the German Medical Device Act (MPG), which includes the national implementation of EC directive 93/42/EEC.

DETAILED DESCRIPTION:
The aim of this non-randomized post-market clinical follow-up study is to confirm long-term safety and effectiveness of the CE-approved Camouflage-coated self expandable RESISTANT Camouflage stent system for revascularization of de novo stenotic lesions in superficial femoral artery in 120 compliant patients suitable for stent angioplasty. The primary end point is the target lesion revascularization after 12 months. Further follow-ups are scheduled at discharge, 30 days, 6 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 95 years
* Male or non-pregnant female
* De novo lesions>70% or occlusions in the SFA (Superficial Femoral Artery) arteries suitable for stent angioplasty
* Max. 1 lesion within each leg should be treated as study lesions
* Lesions length range from ≥3 cm to ≤18 cm
* A patent inflow artery free from significant lesions (>50 % stenosis) as confirmed by angiography. Treatment of target lesion acceptable after successful treatment of inflow artery lesions.
* Reference vessel diameter ≥3 mm and ≤ 7 mm
* Successful guide wire passage of the lesion
* Symptomatic peripheral artery disease (Rutherford stage 2 to 5)
* Patient is willing to provide informed consent and comply with the required follow-up visits, testing schedule, and medication regimen

Exclusion Criteria:

* Patients for whom an anti-platelet therapy, anticoagulants or thrombolytics are contraindicated
* Patients presenting a lasting intraluminal thrombosis at the lesion after a thrombolytic therapy
* Perforation at the location of the angioplasty characterized by secretion of the contrast medium
* Aneurysm of the artery to be treated
* All common contraindications for a PTA (Percutaneous Transluminal Angioplasty)
* Contraindications for stent angioplasty
* Hypersensitivity/allergy to nickel-titanium
* Hypersensitivity/allergy to any of the components of the delivery & dilation system
* Severe renal insufficiency (creatinine>2.0 mg/dL or glomerular filtration rate < 60 ml/min/1.73)
* Uncorrected bleeding disorder
* Major gastrointestinal bleeding within the last 6 months.
* Ipsilateral intervention other than target vessel
* Untreated ipsilateral iliac artery stenosis >70 %
* Previous stenting or prior surgery of the SFA
* In-stent restenosis
* Acute myocardial infarct within 72 h
* Less than one patent crural artery
* Popliteal stenosis > 70 %
* Manifest hyperthyroidism
* Acute onset of symptoms
* Leg-threatening ischemia
* Multimorbid patient with poor general condition
* Pregnant woman or becoming pregnant in < 2 yrs
* Living more than 100 km apart from the study center
* Patient actively participating in another investigational device or drug study
* History of hemorrhagic stroke within 3 months
* Previous or planned surgical or interventional procedure within 30 days of the procedure
* Acute or sub-acute thrombus in target vessel
* Acute vessel occlusion or sudden symptom onset
* Lesions in target area requiring atherectomy (or ablative devices), cutting balloons, cryoplasty balloons, or any other advanced device to facilitate angioplasty balloon or stent delivery
* Use of adjunctive therapies (i.e. laser, atherectomy, cryoplasty, scoring/cutting balloon, etc.)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with de novo stenotic lesions in the superficial femoral artery
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-03 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Target lesion revascularization (TLR) | 12 months
  Target lesion revascularization (TLR) rate

SECONDARY OUTCOMES:
Adverse Event | 24 hours
  Adverse Event rate
Adverse Event | 48 hours
  Adverse Event rate
Adverse Event | 6 months
  Adverse Event rate
Adverse Event | 12 months
  Adverse Event rate
Adverse Event | 24 months
  Adverse Event rate
Technical success | 24 hours
  The ability to successfully complete stent angioplasty and achieve a residual diameter stenosis of ≤ 30 %.
Procedural success | 24 hours
  Procedural success rate
Walking Impairment Questionnaire | 6 months
  Change from baseline in Walking Impairment Questionnaire scores
Walking Impairment Questionnaire | 12 months
  Change from baseline in Walking Impairment Questionnaire scores
Rutherford classification | 48 hours
  Change from baseline in Rutherford stage
Rutherford classification | 6 months
  Change from baseline in Rutherford stage
Rutherford classification | 12 months
  Change from baseline in Rutherford stage
Rutherford classification | 24 months
  Change from baseline in Rutherford stage
Health-related quality of life (SF-36 questionnaire) | 12 months
  Change from baseline in health-related quality of life (SF-36 questionnaire scores)
Primary patency | 6 months
  Percentage of lesions that reach endpoint without TLR or with stenosis < 50% on duplex ultrasonography (PSVR (Peak Systolic Velocity Ratio) < 2.4)
Primary patency | 12 months
  Percentage of lesions that reach endpoint without TLR or with stenosis < 50% on duplex ultrasonography (PSVR (Peak Systolic Velocity Ratio) < 2.4)
Primary patency | 24 months
  Percentage of lesions that reach endpoint without TLR or with stenosis < 50% on duplex ultrasonography (PSVR (Peak Systolic Velocity Ratio) < 2.4)
Ankle brachial index (ABI) | 48 hours
  Change from baseline in Ankle brachial index (ABI)
Ankle brachial index (ABI) | 6 months
  Change from baseline in Ankle brachial index (ABI)
Ankle brachial index (ABI) | 12 months
  Change from baseline in Ankle brachial index (ABI)
Ankle brachial index (ABI) | 24 months
  Change from baseline in Ankle brachial index (ABI)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Giese, Phd, Study Chair — Eucatech AG
Locations (5):
- Germany (4):
  - Uniklinikum Freiburg, Abteilung Röntgendiagnostik, Freiburg im Breisgau, Baden-Wurttemberg
  - Uniklinikum Gießen und Marburg, Diagnostische und Interventionelle Radiologie, Marburg, Hesse
  - Augusta-Krankenhaus, Klinik für Gefäßchrirugie, Düsseldorf, North Rhine-Westphalia
  - Heinrich Braun Klinikum Zwickau, Radiologie und Neuroradiologie, Zwickau, Saxony
- CCP - Istituto di Cura "Città di Pavia", Pavia, Lombardy, Italy